Neurosciences Building Department of Psychiatry Warneford Hospital Warneford Lane OX3 7JX Oxford



Professor Philip J Cowen Principal Investigator 01865 618311 phil.cowen@psych.ox.ac.uk

Doctor Riccardo De Giorgi Graduate reading for DPhil in Biomedical and Clinical Sciences 01865 618238 riccardo.degiorgi@bnc.ox.ac.uk

## PARTICIPANT CONSENT FORM

MS IDREC Approval Reference: R61966/RE001

## The effect of seven-day atorvastatin administration on emotional processing, reward processing, and inflammation in healthy volunteers

Purpose of Study: To investigate the effect of seven-day atorvastatin administration on emotional processing, reward processing, and inflammation.

| | | Please initial each<br>box |
|---|---|---|
| 1 | I confirm that I have read and understand the information sheet version 1.0 dated 01 <sup>st</sup> January 2019 for the above study. I have had the opportunity to consider the information carefully, ask questions and have had these questions answered satisfactorily. | |
| 2 | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, and without any adverse consequences or academic penalty. | |
| 3 | I have been advised about the potential risks associated with taking part in this research and have taken these into consideration before consenting to participate. | |
| 4 | I have been advised as to what I need to do for this research (especially with regard to drug intake) and I agree to follow the instructions given to me. | |
| 5 | To the best of my knowledge, I do not meet any of the exclusion criteria outlined in the information sheet for this research. If this changes at a later date during study participation, I agree to notify the researchers immediately. | |
| 6 | I understand that data collected during the study may be looked at by designated individuals from the University of Oxford. I give permission for these individuals to access my data. | |
| 8 | I understand who will have access to personal data provided, how the data will be stored, and what will happen to the data at the end of the project. | |
| 9 | I agree for data collected in this study to be shared with other researchers, including those working outside of the EU, to be used in other research studies. I understand that any data shared will be fully anonymised so that I cannot be identified. | |

| Name of r | person taking consent | dd / mm / yyyy<br>Date | <br>Signature |
|---|---|---|---|
| Name of p | participant | Date | Signature |
| | | dd / mm / yyyy | |
| Optional: | contacting me about futur | details to be kept in a secure database for the purpose of future studies. I understand that agreeing to be contacted participate in any further studies. | |
| 13 | | | |
| 12 | I agree to take part in the study | | |
| 12 | understand how to raise a concern or make a complaint. | | |
| 11 | I understand that this project has been reviewed by, and received ethics clearance through, the University of Oxford Central University Research Ethics Committee. | | |
| 10 | I understand how this rese | earch will be written up a | and published. |